CLINICAL TRIAL: NCT04913961
Title: Efficacy Evaluation of Supine Daoyin in the Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease: A Multi-center, Randomized Controlled Trial
Brief Title: Supine Daoyin in the Treatment of AECOPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Daoyin for AECOPD
Record Dates: First submitted 2021-04-26; First posted 2021-06-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Acute exacerbation; Pulmonary rehabilitation; Supine Daoyin; Randomized controlled trail
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine Daoyin (Experimental): During hospitalization, the rehabilitation group will receive conventional western medicine treatment and supine guidance therapy which consists of training and patient education. They will be evaluated with some tests for the study.
  Interventions: Other: Supine Daoyin
- Control (Active Comparator): The control group will get the western medicine conventional therapy with some additional tests for the study.
  Interventions: Other: western medicine conventional therapy

INTERVENTIONS:
Other: Supine Daoyin — During hospitalization, the rehabilitation group will receive conventional western medicine treatment and supine guidance therapy which consists of training and patient education. They will be evaluated with some tests for the study
  Arms: Supine Daoyin
Other: western medicine conventional therapy — The control group will get the western medicine conventional therapy with some additional tests for the study.
  Arms: Control

SUMMARY:
The purpose of this study was to evaluate the clinical efficacy and safety of supine daoyin in the treatment of AECOPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a chronic progressive disease with high incidence rate, high mortality rate and high disability rate. Among the people over 40, the prevalence rate is 10.1%, while the prevalence rate in China is 13.7%. Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) is a major event that affects the natural course of COPD. In particular, most patients with AECOPD have poor prognosis, higher morbidity and mortality, and lower quality of life. Pulmonary rehabilitation can improve the clinical symptoms of AECOPD patients, increase exercise tolerance, delay the decline of lung function, and improve the quality of life. In recent years, the clinical research on the rehabilitation of patients with AECOPD is still in the exploratory stage, which needs to be supported by clear evidence.

This is a multicenter, randomized controlled trial to evaluate the clinical efficacy and safety of supine daoyin in the treatment of AECOPD. After admission, the patients were randomly divided into two groups, rehabilitation group and control group, 114 cases in each group. After routine treatment, the patients began to recover when they reached the initial rehabilitation standard, and recovered until they reached the discharge standard. The primary outcomes are the length of hospital stay due to acute exacerbation and clinical symptom score. The secondary outcomes include activities of daily living, dyspnea score, 6-minute walking distance, lower limb muscle strength, mechanical ventilation and quality of life. Safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of AECOPD.
2. Age between 40 and 80 years.
3. mMRC score ≥ 3.
4. Barthel index<50.
5. With the informed consent signed.

Exclusion Criteria:

1. Patients with severe cognitive impairment, dementia and various psychosis.
2. Combined with severe arthritis and other osteoarthritis affecting the movement.
3. Dyskinesia due to neuromuscular diseases.
4. Long term bedridden for various reasons.
5. Participating in other trials.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay due to acute exacerbation | through study completion, an average of 2 weeks
  The time from hospitalization to discharge was counted
Clinical symptom assessment questionnaire (CCQ) | Change from baseline CCQ scores at day 3，day 7，day 14
  The Clinical symptom assessment questionnaire (CCQ) is a self-administered questionnaire that measures health-related quality of life. It is an 10-item questionnaire on a 0-6 point scale with higher values indicating greater impact of COPD.

SECONDARY OUTCOMES:
Activities of daily living (Barthel index) | Change from baseline Barthel index scores at day 3，day 7，day 14
  Activities of daily living (ADL): the scale includes 10 items, including 8 items of self-care activities and 2 items of action related activities, with a total score of 100.
Borg dyspnea score | Change from baseline Borg dyspnea score at day 3，day 7，day 14
  Borg dyspnea score is is a 10-point (0-10) scale based on the severity of dyspnoea. "0" means no dyspnea perception, "10" means most severe dyspnea perception.
30-second sit-to-stand test | Change from baseline 30-second sit-to-stand test at day 3，day 7，day 14
  Record the times of sitting and standing test within 30 seconds
Mechanical ventilation | through study completion, an average of 2 weeks
  The number of patients using noninvasive or invasive mechanical ventilation during the study period was counted
6 Minutes Walking Distance Test (6MWD) | Change from baseline 6MWD test at day 7，day 14
  The 6-minute walking distance of the two groups was calculated
St. George's Respiratory Questionnaire（SGRQ） | Change from baseline SGRQ scores at day 3，day 7，day 14
  The St. George's Respiratory Questionnaire (SGRQ) scores will be used to evaluate quality of life with a total score of 0-100. The higher scores will indicate the worse outcomes.
The modified COPD Patient-Reported Outcome scale (mCOPD-PRO) | Change from baseline mPRO-COPD scores at day 3，day 7，day 14
  The modified COPD Patient-Reported Outcome scale (mCOPD-PRO) will be used to assess quality of life. The mCOPD-PRO contains 27 items in three domains. mCOPD-PRO scores range from 0 to 4 with a decrease in score showing higher health status.
The modified Effectiveness Satisfaction Questionnaire for COPD (mESQ-COPD) | Change from baseline mESQ-COPD scores at day 3，day 7，day 14
  The modified Effectiveness Satisfaction Questionnaire for COPD (mESQ-COPD) will be used to assess treatment satisfaction. The mESQ-COPD contains 19 items in four domains. mESQ-COPD scores range from 0 to 4 with a decrease in score showing higher treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Li jiansheng, doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Chinese, Zhengzhou, Henan, China